CLINICAL TRIAL: NCT03173079
Title: Geriatric Assessment and Outcome in Patients Undergoing Transcatheter Aortic Valve Replacement
Status: Completed | Type: Observational
Sponsor: Campus Bad Neustadt (Other)
Collaborators: Rhönklinikum AG (Unknown)
Responsible Party: Principal Investigator, Sebastian Barth, PI, Campus Bad Neustadt
Other Study IDs: CampusBN
Record Dates: First submitted 2017-05-30; First posted 2017-06-01 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Influence of Geriatric Functional State on the Outcome After TAVI; Possible Change in Geriatric Assessment After TAVI
MeSH Terms: interventions — Lead

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: pre- and postinterventional geriatric assessment in patients undergoing TAVI — geriatric assessment

SUMMARY:
A geriatric assessment is becoming increasingly important in the treatment of patients with a percutaneous aortic valve replacement due to their comorbidities. The aim of this multimodal therapy concept is to examine the influence on the postoperative outcome. In addition to a comprehensive assessment of the individual frailty score, the subjective condition before and after TAVI is also evaluated using a standardized questionnaire ("Minnesota living with heart failure questionnaire").

ELIGIBILITY:
Inclusion Criteria:

* all patients with indication for TAVI according to the current guidelines

Exclusion Criteria:

* no indication for TAVI, indication for cardiac surgery, mentally disabled patients, patients with endocarditis or life expectancy of less than 2 years

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: all-comers cohort
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
Quality of Live score in the "Minnesota living with heart failure questionnaire" | 6 month
  self reported quality of life
frailty score | 6 month
  multimodal geriatric assessment including cognitive Status (MMST, clock test, Tinetti test, stand up and go-test)
mortality after TAVI | 6 month
  phone call follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Barth, MD, Principal Investigator — Cardiovascular Center Bad Neustadt; Karsten Hamm, MD, Principal Investigator — Cardiovascular Center Bad Neustadt
Locations (1):
- Cardiovascular Center Bad Neustadt, Bad Neustadt an der Saale, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Undecided